CLINICAL TRIAL: NCT06725329
Title: Developing a Tailored Psychosocial Education Intervention for Chronic Pain Management for Asian Americans in the Community
Brief Title: Developing a Tailored Psychosocial Education Intervention for Chronic Pain Management for Asian Americans
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Hee Jun Kim, Associate Professor, George Washington University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCR235347; 1R21NR021224-01 (NIH)
Record Dates: First submitted 2024-11-15; First posted 2024-12-10 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Chronic Pain
Keywords: tailored psychosocial education intervention; pain disparity; korean Americans; Asian Americans; Chronic Pain; Learn About My Pain(LAMP) program; Pain intensity; Pain interference; Pain catastrophizing; community-based pain management program; culturally adapted
MeSH Terms: conditions — Chronic Pain; Pain

STUDY DESIGN:
Intervention Model Description: The investigators will use a three-phase integrated sequential approach (Qual-Quant-Qual). The first stage is a qualitative phase to adapt and culturally-integrate the psychosocial intervention for KA. Focus group discussions (FGDs) with individuals with lived experience (n = 15) will be conducted in KA. Upon analysis of the FGDs with study participants, the findings will be used to adapt a previously developed psychosocial education intervention for KA (Aim 1). The second phase involves pilot testing the tailored intervention using a single-group, pre-posttest design (n = 30). The last stage will involve post intervention individual, semi-structured in-depth interviews that will focus on participants' reflections of the sessions in relevance to their culture and pain management (n = 10). The feasibility and acceptability of the tailored intervention will be assessed by integrating the qualitative and quantitative findings (Aim 2).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adapted and culturally-integrated psychosocial education intervention (Experimental): Participants will receive the culturally adapted psychosocial educational program for chronic pain management. The investigators will adapt the Learn About My Pain (LAMP) program that has previously been established for efficacy in reducing chronic pain intensity, pain interference, and pain catastrophizing in racialized groups in community settings. The LAMP intervention provides biopsychosocial education sessions about chronic pain and its management.
  Interventions: Behavioral: A tailored psychosocial education intervention

INTERVENTIONS:
Behavioral: A tailored psychosocial education intervention — Participants will get ten 60-minute psychoeducational group sessions about chronic pain and its management. The group sessions will be conducted by the PI and a bilingual project director at Korean churches or daycare centers in Baltimore-Washington Metropolitan area.
  The psychoeducational group session will be adapted from LAMP intervention that has been previously developed. The intervention provides biopsychosocial education sessions about chronic pain and its management. For example, sessions focus on providing information regarding: (1) pain and the biological stress response and the gate control theory of pain, (2) the psychological impact of thoughts and emotions on pain and (3) facilitated group discussions to help participants develop a new understanding of pain through shared social experiences, all of which have been shown to improve pain outcomes.

SUMMARY:
Health inequalities in chronic pain exists in the US, with a greater burden of chronic pain and higher rate of misdiagnosis and undertreatment reported in minoritized groups compared to non-Hispanic Whites. Asian Americans (AA) are the fastest-growing racial/ethnic group in the US, yet despite the rapid growth in their numbers, AA remain under-represented in pain disparity research. Cultural norms of Asians may discourage reporting their pain to avoid burdening others or being seen as weak. Rather than seeking medical assistance, Asians have been reported to tend to accept the pain as natural or to suffer to maintain their independence. Very few evidence-based programs are available that can be implemented for this linguistically/socially isolated population in the US. This proposed study aims to fill critical knowledge gaps in pain disparity research by providing evidence of feasibility and acceptability of a culturally-tailored psychosocial pain education intervention for an underrepresented population using the KA community as an exemplar.

DETAILED DESCRIPTION:
Chronic pain is a major population health issue affecting more than 100 million Americans and disparities in chronic pain have been widely documented, indicating minoritized racial and ethnic groups experience a higher burden of chronic pain and are at high risk for undertreatment of that pain. Asian Americans remain underrepresented in pain research; evidence regarding chronic pain experiences of Asian Americans is limited, as are resources and evidence-based programs for this group. This exploratory, developmental study will provide evidence of feasibility and acceptability of a culturally tailored psychosocial education intervention to reduce pain catastrophizing and improve pain outcomes for underrepresented and underserved minority populations.

ELIGIBILITY:
Inclusion Criteria:

1. Female and male
2. ≥ 18 years old
3. Self-reported foreign born Korean Americans
4. Self-reported pain most days of the month for at least 3 months
5. Pain must be non-malignant, but may have more than one pain source

Exclusion Criteria:

1. Having malignant pain (e.g., cancer or HIV-related)
2. Demonstrating significant cognitive impairment (based on results of a cognitive screener-Short Portable Mental Status Questionnaire)
3. Having current, uncontrolled serious psychological disturbance (e.g., schizophrenia, bipolar disorder) or active substance abuse based on self-report
4. Having low literacy skills in Korean or English (unable to understand the written consent and to sign)
5. Undergoing other psychosocial treatment for pain

   * If excluding a population or group that may benefit from the research, please provide justification: We will exclude children. The original intervention (LAMP) trial has established for efficacy in reducing chronic pain outcomes in adult population. Children are not our target population as we focus on developing a culturally tailored chronic pain management program based on LAMP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-03-08 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility_Recruitment/retention | From T1 (enrollment) to T2 (at completion of the 10 week session)
  Recruitment rates will be monitored over the recruitment periods, and reasons for non-consent will be recorded. Retention will be monitored across T1 to T2, and if participants withdraw during the study periods, they will be asked for reasons and invited to the post-intervention interviews to elaborate on their choice to withdraw.
Pain Outcomes_Pain Catastrophizing | T1 (enrollment), T2 (after the 10 week sessions), and T3(Twelve weeks after the intervention)
  Pain catastrophizing will be measured using the Pain Catastrophizing Scale (PCS), a 13-item scale that assesses catastrophic thinking, including subscales of helplessness, rumination, and magnification, in response to pain. The PCS total score will be calculated by summing the total item responses; higher scores on the PCS are indicative of greater pain-related catastrophizing.
Pain Outcomes_Pain Interference | T1 (enrollment), T2 (after the 10 week sessions), and T3(Twelve weeks after the intervention)
  Pain interference will be also measured using the BPI-SF subscale. The subscale evaluates the degree of interference with general activity, mood, walking, work, sleep, relations with using a numeric rating scale (0 = 'no interference' and 10 = 'interferes completely).
Pain Outcomes_Pain Intensity | T1 (enrollment), T2 (after the 10 week sessions), and T3(Twelve weeks after the intervention)
  Pain intensity will be measured using the 4-item Brief Pain Inventory-Short Form (BPI-SF) Pain Intensity subscale, which uses an 11-point numeric rating scale (0 = 'no pain' and 10 = 'pain as bad as you can imagine') to evaluate pain at its worst, least, average, and current severity over the past week.
Feasibility_Participant engagement | 4 Week, 8 Week, T2(10 Week)
  Participant engagement will be tested by the number of completed sessions, including completion of weekly activities (i.e., coping strategies).
Feasibility_Participant satisfaction | 4 Week, 8 Week, T2(10 Week)
  Participant satisfaction will be measured by one item asking, "Overall, how satisfied were you with the 10 -week pain management program?" The item will be rated on a 7-point Likert scale from very dissatisfied to very satisfied.
Feasibility_Barriers/facilitators to engagement | Within 2 weeks upon the completion of the final session(10-12 Week)
  Individual, semi-structured in-depth interviews will be conducted within 2 weeks upon the completion of the final session to obtain participants' reflections of and feedback on the program.
Acceptability_Perceived appropriateness | Within 2 weeks upon the completion of the final session(10-12 Week)
  Individual, semi-structured in-depth interviews will be conducted within 2 weeks upon the completion of the final session to obtain participants' reflections of and feedback on the program.
  Acceptability is defined as the perception that a new intervention is agreeable or satisfactory. Perceived appropriateness for the intervention format, the lengths of the group session, and the total intervention program will be assessed using semi-structured interviews with subset of study participants (n = 10).

SECONDARY OUTCOMES:
Health status (Physical/mental well-being) | From Enrollment (T1), Week 10 (T2), Week 22 (T3)
  Health status will be measured using the Short Form (SF)-12 to capture physical and mental well-being and limitations. The SF-12 score is a measure of both physical and mental well-being, with a higher score indicating better overall health, where scores are typically interpreted with a range of 0-100, with a score above 50 generally considered to be within a healthy range for both physical and mental components; the SF-12 calculates separate "Physical Component Summary (PCS)" and "Mental Component Summary (MCS)" scores based on responses to 12 questions covering different aspects of health like physical functioning, bodily pain, vitality, and mental health.
  The SF-12 assesses eight health domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. The Korean version of the SF-12 v2 that has been previously validated will be used for this study.
Acculturation | Enrollment (T1)
  Acculturation will be measured using the Short Acculturation Scale, which includes 12 items focusing on language use, media use, and ethnic social relations
Social Isolation | Enrollment (T1)
  Social Network will be assessed by using the Lubben Social Network Scale to measure contacts, talks, and supports from family and friends networks.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - The George washington University, Washington D.C., District of Columbia
  - George Washington University School of Nursing, Ashburn, Virginia

IPD SHARING:
Plan to Share IPD: Undecided
The research team has not decided whether the IPD will or not be shared. The research team will discuss this matter after the trial is completed.